CLINICAL TRIAL: NCT07292337
Title: Pain Relief by Applying Transcutaneous Electrical Nerve Stimulation (TENS) During Transrectal Ultrasound Guided (TRUS) Prostate Biopsy: A Randomized Double-blind Placebo-controlled Trial
Brief Title: AcuTENS for Pain Relief During TRUS-Guided Prostate Biopsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Harshini Mahendran, Research Team member, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UMG012C-2024; UMG012C-2024 (Other Grant/Funding Number: Mahmood Merican Research Grant, University of Malaya)
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Procedural Pain Relief; TRANSRECTAL ULTRASOUND-GUIDED PROSTATE BIOPSY; Transcutaneous Electrical Nerve Stimulation
Keywords: Transcutaneous electrical nerve stimulation; TRUS-guided prostate biopsy; Pain control and anxiety management during procedure
MeSH Terms: conditions — Prostatic Neoplasms; Agnosia

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 parallel-group design comparing interventional group using active AcuTENS with placebo TENS during TRUS-guided prostate biopsy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and all study personnel, including clinicians performing the biopsy and assessors recording outcomes, are blinded to group allocation. Intervention devices are identical in appearance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active AcuTENS (Experimental): Participants receive active transcutaneous electrical nerve stimulation applied to selected acupuncture points before and during TRUS-guided prostate biopsy, in addition to standard periprostatic nerve block.
  Interventions: Device: Active AcuTENS
- Placebo TENS (Placebo Comparator): Participants receive a identical TENS device with a placebo setting and no therapeutic electrical output, applied to the same acupuncture points before and during TRUS-guided prostate biopsy, in addition to standard periprostatic nerve block.
  Interventions: Device: Placebo TENS

INTERVENTIONS:
Device: Active AcuTENS — Electrical stimulation delivered via surface electrodes placed on predefined acupuncture points. Stimulation is applied before and during the biopsy using a device capable of therapeutic current output.
  Arms: Active AcuTENS
Device: Placebo TENS — An identical TENS device set to a placebo setting with no active electrical output. Electrodes are applied to the same acupuncture points, with no therapeutic stimulation.
  Arms: Placebo TENS

SUMMARY:
This study evaluates whether transcutaneous electrical nerve stimulation applied at specific acupuncture points (AcuTENS) can reduce pain and anxiety during transrectal ultrasound-guided prostate biopsy for participants suspected of prostate cancer. Many patients experience significant discomfort despite the use of periprostatic nerve block (PPNB).

The aim of this study is to determine whether AcuTENS provides additional pain relief or anxiety reduction beyond standard analgesia. The findings may help identify a simple, low-risk adjunct that can improve patient comfort during prostate biopsy. AcuTENS is a non-invasive technique that delivers mild electrical stimulation through the skin, targeting acupuncture points believed to modulate pain perception.

In this randomized, double-blind, placebo-controlled trial, participants are assigned to receive either active AcuTENS or a placebo TENS device that produces no therapeutic stimulation . All participants with receive routine care, including PPNB, according to institutional protocol. Pain scores, anxiety levels, vital signs, and patient satisfaction are recorded before, during, and after the biopsy.

DETAILED DESCRIPTION:
Transrectal ultrasound-guided prostate biopsy is the standard diagnostic procedure for suspected prostate cancer. Despite routine analgesic strategies such as periprostatic nerve block, many patients continue to experience moderate pain and procedure-related anxiety.

AcuTENS, a form of transcutaneous electrical nerve stimulation applied to acupuncture points, has shown potential benefits in chronic pain conditions, osteoarthritis, and procedural discomfort in small-scale studies. Its proposed mechanism involves activation of peripheral nerve fibers, endogenous opioid pathways, and autonomic modulation, leading to reduced pain perception and improved relaxation. However, high-quality randomized controlled data for its use during prostate biopsy are limited.

This study is a randomized, double-blind, placebo-controlled clinical trial conducted at University Malaya Medical Centre. The trial consists of two arms:

1. Active AcuTENS: Electrical stimulation applied to predetermined acupuncture points before and during the biopsy.
2. Placebo TENS: Identical device with no therapeutic electrical output.

An initial pilot phase involving 10 patients demonstrated that AcuTENS was feasible, safe, and potentially beneficial. This informed the development of the current definitive trial, which includes 53 participants.

All participants undergo the standard TRUS-guided prostate biopsy with local anesthesia using PPNB. Pain (VAS), anxiety (standardized scales), heart rate, blood pressure, and patient satisfaction are assessed at predefined time points.

The primary outcome is assessment of pain during insertion of ultrasound probe, injection of local anaesthesia and pain during collection of biopsy. Secondary outcomes include anxiety reduction, hemodynamic stability, satisfaction scores, and any adverse effects related to TENS use.

This investigation aims to determine whether AcuTENS offers meaningful improvement in patient comfort during prostate biopsy. If effective, it could be incorporated into routine practice as a simple, safe, and affordable adjunct to existing analgesic measures.

ELIGIBILITY:
Inclusion Criteria:

1. Patient consented for first time TRUS prostate biopsy.
2. Patient aged 18 years and above.

Exclusion Criteria:

1. Patient with previous experience of TRUS biopsy
2. Patient with pacemakers or automatic cardiac defibrillator implant or implant in the upper limb
3. Patient with cutaneous skin breaks on application sites (e.g wound, burn scar)
4. Patient diagnosed to have epilepsy or impaired mental state or anxiety disorder
5. Patient with known allergy to acupuncture patch or lidocaine spray

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy pain relief of application of Acu-TENS in TRUS prostate biopsy | VAS scores will be recorded in real time at the moment of maximal discomfort during: Insertion of the transrectal ultrasound probe Injection of periprostatic local anaesthesia Prostate biopsy sampling Time Frame: Immediately during the procedure
  Pain intensity will be assessed using the Visual Analogue Scale (VAS), a validated pain measurement tool ranging from 0 to 10, where:
  0 = no pain 10 = worst pain imaginable Higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
To evaluate anxiety levels of subjects undergoing TRUS biopsy with application of Acu-TENS | STAI scores will be measured: 1. Before the biopsy 2. Immediately after completion of the biopsy Time Frame: Pre-procedure and immediately post-procedure
  Anxiety will be assessed using the State-Trait Anxiety Inventory (STAI), a validated self-reported questionnaire consisting of two subscales:
  State Anxiety (STAI-S): measures situational anxiety at a specific time Trait Anxiety (STAI-T): measures baseline anxiety tendency
  Each subscale score ranges from 20 to 80, with:
  Lower scores indicating lower anxiety Higher scores indicating greater anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Dr Novinth Kumar A/L Raja Ram, MBBS, MS (Gen Surg), Principal Investigator — Department of Surgery (Urology Unit), University Malaya Medical Centre, Kuala Lumpur, Malaysia
Locations (1):
- University of Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nazir B. Pain during transrectal ultrasound-guided prostate biopsy and the role of periprostatic nerve block: what radiologists should know. Korean J Radiol. 2014 Sep-Oct;15(5):543-53. doi: 10.3348/kjr.2014.15.5.543. Epub 2014 Sep 12. PMID 25246816
- [Result] Ouzounidis X, Moysidis K, Kalinderis N, Papanikolaou D, Koukourikis P, Papaefstathiou E, Hatzimouratidis K. Efficacy and safety of three different analgesic methods for patients undergoing transrectal ultrasound-guided prostate biopsy: a prospective, randomized controlled trial. Hippokratia. 2020 Oct-Dec;24(4):166-172. PMID 35023892
- See also: Pain as the 5th Vital Sign Guideline — https://www.moh.gov.my/moh/resources/Penerbitan/Program%20Bebas%20Kesakitan/Garis%20Panduan/2_in_1_P5VS_Guideline_3rd_Edition_Corrected_2020.pdf